CLINICAL TRIAL: NCT06560671
Title: Compare the Patient Satisfaction and Effectiveness After Novel Application-based or Conventional Health Education of Bowel Preparation for Colonoscopy-- Randomized Controlled Trial
Brief Title: Compare the Patient Satisfaction and Effectiveness After Novel Application-based or Conventional Health Education of Bowel Preparation for Colonoscopy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 202310047RINB
Record Dates: First submitted 2024-08-11; First posted 2024-08-19 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Colo-rectal Cancer; Colon Lesion
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional (Other)
  Interventions: Other: novel type of health education
- Novel (Experimental)
  Interventions: Other: novel type of health education

INTERVENTIONS:
Other: novel type of health education — animation video based health education

SUMMARY:
Colorectal cancer is the cancer with highest incidence in Taiwan. The disease itself and subsequent treatment cause huge impact on the physical, psychological, and spiritual parts and social role of a patient. Early diagnosis of colorectal cancer and precancerous lesions is possible. Early treatment can reduce the impact on quality of life and economics.

Colonoscopy is an important tool for diagnosis of colorectal proliferative lesions. Qualified bowel preparation can enhance sensitivity and reduce false negative of the colonoscopy. However, multiple factors influence the quality of bowel preparation. This study aims to investigate whether the animation video and game-based health education is more effective and satisfying than conventional health education, and to explore the difference of knowledge dissemination and quality of bowel preparation between novel and conventional methods.

This study is a randomized controlled trial and uses structural questionnaire for study participants. Before the main study, the investigators will consult professors' opinions to adjust and enhance validity of the questionnaire, and the investigators will perform pretest to calculate its reliability. The investigators will enroll participants at the out-patient-department and the health management center. Questionnaires may be completed by on-site paper or phone with internet resources. The main participants of this study are adults aged 18 and more, and planned to receive colonoscopy. The questionnaires investigate the spent time, patient satisfaction, knowledge of bowel preparation and results of colonoscopy of different approaches of health education. Multiple linear regression will be applied to calculate the possible significance difference between two kinds of health education.

The investigators expect this study (1) to explore whether novel health education enhances patient satisfaction (2) to investigate the efficiency of novel health education, and (3) to compare the effect of knowledge dissemination and quality of bowel preparation between experimental and control groups. This study will develop the model of health education to facilitate holistic health care.

ELIGIBILITY:
Inclusion Criteria:

* adults planned to accept colonoscopy exam

Exclusion Criteria:

* can't accept health education or refuse follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
quality of bowel preparation | immediately after the procedure of colonoscopy
  cleansing level of Aronchick scale 1-4

SECONDARY OUTCOMES:
satisfaction of health education | immediately after the intervention of health education
  5 points Likert scale

CONTACTS AND LOCATIONS:
Overall Officials: Mingchih Liu, MD, Principal Investigator — National Taiwan University Hospital Hsinchu Branch
Locations (1):
- National Taiwan University Hsinchu Branch, Hsinchu, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided